CLINICAL TRIAL: NCT02848365
Title: Incidence and Severity of Postoperative Sore Throat And Intubation Response by Using Different Devices for Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Mansoor Aqil, Professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: E-11-398
Record Dates: First submitted 2016-07-22; First posted 2016-07-28 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Pharyngitis; Endotracheal Intubation; Pain
Keywords: Measurement
MeSH Terms: conditions — Pharyngitis; Pain | interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- Glidescope (Active Comparator)
  Interventions: Device: Endotracheal intubation
- Macintosh laryngoscope (Active Comparator)
  Interventions: Device: Endotracheal intubation
- Bonfill's rigid scope (Active Comparator)
  Interventions: Device: Endotracheal intubation
- Air traq (Active Comparator)
  Interventions: Device: Endotracheal intubation
- C -Mac scope (Active Comparator)
  Interventions: Device: Endotracheal intubation
- flexible fiberoptic scope (Active Comparator)
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: Endotracheal intubation — Endotracheal intubation will be done with any of these equipments

SUMMARY:
Postoperative sore throat (POST) is a common problem following the use of endotracheal intubation during general anaesthesia. It leads to dissatisfaction and discomfort after surgery and can delay a patient's return to normal routine activities. POST has been rated by patients as the eighth most adverse effect in the postoperative period. The incidence of sore throat after endotracheal intubation varies from 14.4-90%. Laryngoscopy and tracheal intubation also leads to hemodynamic stress response. The response can be deleterious in patient with or without cardiac disease. It is related to the degree of manipulation of the airway during endotracheal intubation and has been studied during intubation for some equipment used for endotracheal intubation

ELIGIBILITY:
Inclusion Criteria:

* After signing of the informed consent,
* ASA physical status I and II
* Mallampati class 1& 2,
* BMI < 35,
* Undergoing elective surgical procedures (not exceeding two hours in duration) requiring ET intubation

Exclusion Criteria:

* Patients undergoing day case,
* bariatric, cardiac, nasal, oral or head & neck surgeries,
* requiring placement of throat pack or nasogastric/ orogastric tube,
* patients assigned to rapid sequence induction,
* hoarseness,
* patients with anticipated difficult intubation,
* history of recent upper respiratory tract infection,
* history of difficult intubation
* psychiatric disorders hindering proper evaluation,
* use of steroids (oral or inhalational) or non-steroidal anti-inflammatory drugs within one week of surgery or previous surgery within last two weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2011-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Incidence of post operative sore throat | 0 hours after surgery
Incidence of post operative sore throat | 6 hours after surgery
Incidence of post operative sore throat | 12 hours after surgery
Incidence of post operative sore throat | 24 hours after surgery
Severity of post operative sore throat | 0 hours after surgery
Severity of post operative sore throat | 6 hours after surgery
Severity of post operative sore throat | 12 hours after surgery
Severity of post operative sore throat | 24 hours after surgery
Mean arterial pressure after endotracheal intubation | 1 minute after surgery
Mean arterial pressure after endotracheal intubation | 2 minutes after surgery
Mean arterial pressure after endotracheal intubation | 3 minutes after surgery
Mean arterial pressure after endotracheal intubation | 4 minutes after surgery
Mean arterial pressure after endotracheal intubation | 5 minutes after surgery

SECONDARY OUTCOMES:
cormack Leehanes grade of laryngeal view | At the time of intubation
Percentage of glottic opening score (POGO) score | At the time of intubation
Intubation difficulty score | At the time of intubation
Patient's satisfaction score | After 24 hours of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, King Khalid University Hospital, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Aqil M, Khan MU, Mansoor S, Mansoor S, Khokhar RS, Narejo AS. Incidence and severity of postoperative sore throat: a randomized comparison of Glidescope with Macintosh laryngoscope. BMC Anesthesiol. 2017 Sep 12;17(1):127. doi: 10.1186/s12871-017-0421-4. PMID 28899338